CLINICAL TRIAL: NCT01765452
Title: Multi-center, Randomized, Open Study for Comparison of Efficacy and Safety of Plavix With Astrix and Closone in Patients With Post-Percutaneous Coronary Artery Intervention
Brief Title: Phase IV Study to Compare Efficacy and Safety of Plavix 75mg With Astrix 100mg and Closone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJ_CLO_401
Record Dates: First submitted 2013-01-07; First posted 2013-01-10 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closone (Experimental): 75mg/100mg per day, 8weeks, PO
  Interventions: Drug: Closone
- Plavix with Astrix (Active Comparator): 75mg per day, 8weeks, PO 100mg per day, 8weeks, PO
  Interventions: Drug: Plavix with Astrix

INTERVENTIONS:
Drug: Closone — 75mg/100mg, 8weeks, PO
  Arms: Closone
Drug: Plavix with Astrix — 75mg, 100mg a day, 8weeks, PO
  Arms: Plavix with Astrix

SUMMARY:
The Aim of this study is to prove non-inferiority of Closone to the Combination treatment of Plavix with Astrix.

ELIGIBILITY:
Inclusion Criteria:

* Subjects under a stable condition after Post-Percutaneous Coronary Artery Intervention over three months
* 20~86 years old
* Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

* Subject who did not undergo or failed Drug-Stent Implantation
* Subjects who took an anti-coagulant, anti-thrombotic regularlly( ≥ 2weeks in a month) before the study, or plan to have continuous treatment during the study(Except Aspirin alone or combination of Aspirin and Clopidogrel)
* Subjects with a history of substance or alchol abuse
* Subjects with a history of hypersensitivity to Clopidogrel, Aspirin or other NSAIDS
* Subjects having Aspirin or other NSAIDs-induced Asthma or history
* Subjects with Severe hepatopathy(AST and ALT > 5 times the upper limit of normal)
* Subjects with Severe nephropathy(Cr > 3 times the upper limit of normal)
* Subjects with hemorrhage like gastric ulcer, intracranial hemorrhage etc.
* Subjects with high risk of hemorrhage like blood coagulation disorders, uncontrolled severe hypertension, active bleeding, history of severe bleeding
* subjects who are pregnant, breastfeeding
* Subjects not using medically acceptable birth control
* Subjects who are unsuitable to take the Investigational product due to a medical/mental condition
* Subjects inherently having Galactose malobsorption, Lactase deficiency or Glucose-Galactose malobsorption

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baselinine in P2Y12% inhibition at week 8 | Baseline, week 8

SECONDARY OUTCOMES:
Change from baseline in PRU, ARU at week 8 | Baseline, week 8

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Inje university haeundae paik hospital, Busan
  - Kosin university gospel hospital, Busan
  - Pusan national university hospital, Busan
  - Dongguk University Medical Center, Gyeonggi-do
  - Chungbuk national university hospital, Jungbuk
  - Seoul National University Hospital, Seoul
  - SNU Boramae Medical Center, Seoul